CLINICAL TRIAL: NCT06267066
Title: Fractional Carbon Dioxide Laser: A Novel Therapeutic Option for Lichen Simplex Chronicus: A Randomized Controlled Trial
Brief Title: Fractional Carbon Dioxide Laser: A Novel Therapeutic Option for Lichen Simplex Chronicus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lobna Gamal Alieldin, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-232-2022
Record Dates: First submitted 2024-01-19; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Lichen Simplex Chronicus
Keywords: Lichen Simplex Chronicus; Fractional carbon dioxide laser; Depression; Interleukin 31; Nerve Growth Factor; Substance P
MeSH Terms: conditions — Neurodermatitis; Depression; Hereditary Sensory and Autonomic Neuropathies | interventions — Betamethasone Valerate

STUDY DESIGN:
Intervention Model Description: Sixty patients will be divided randomly through closed envelop technique into 2 groups (Group A and B) each of 30 patients. Group A will be subdivided into 2 groups (1 and 2) each of 15 patients. All LSC lesions will be treated in any patient having multiple lesions.
  Group 1 - A: Patients will receive 3 monthly laser sessions, in addition to the use of topical emollients only once daily in between the sessions.
  Group 2 - A: Patients will receive 3 monthly laser sessions, in addition to topical steroids twice daily and topical emollient once daily in between the sessions.
  Group B: Patients will be prescribed topical steroids twice daily and topical emollient once daily for 3 months.
Who Masked: Outcomes Assessor
Masking Description: Experienced dermatologist blinded to the interventions done will assess the patients' at the end of the treatment period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical Corticosteroids (Active Comparator): Patients will be prescribed topical steroids cream twice daily and topical emollient once daily for 3 months.
  Interventions: Drug: Betamethasone Valerate 0.1% Cream; Drug: Vaseline Topical Product
- Fractional carbon dioxide (Active Comparator): Patients will receive 3 monthly laser sessions, in addition to the use of topical emollients only once daily in between the sessions.
  Interventions: Device: SmartXide® fractional carbon dioxide laser; Drug: Vaseline Topical Product
- Combined topical corticosteroids and Laser (Active Comparator): Patients will receive 3 monthly laser sessions, in addition to topical steroids twice daily and topical emollient once daily in between the sessions.
  Interventions: Drug: Betamethasone Valerate 0.1% Cream; Device: SmartXide® fractional carbon dioxide laser; Drug: Vaseline Topical Product

INTERVENTIONS:
Drug: Betamethasone Valerate 0.1% Cream — Moderate potency
  Arms: Combined topical corticosteroids and Laser; Topical Corticosteroids
Device: SmartXide® fractional carbon dioxide laser — Ablative
  Arms: Combined topical corticosteroids and Laser; Fractional carbon dioxide
Drug: Vaseline Topical Product — Emollient

SUMMARY:
The goal of this randomized control trial is to compare the use of fractional carbon dioxide (Co2) laser to topical corticosteroids to treat lichen simplex chronicus (LSC) patients presenting to Dermatology outpatient clinic, Faculty of Medicine, Cairo University.

Participants will:

* Be assessed clinically by doctor
* Biopsies will be taken from them by doctor
* Receive treatment as laser or topical steroids or both
* Fill in depression questionnaire.

Researchers will divide and compare groups as follows:

Sixty patients will be divided randomly through closed envelop technique into 2 groups (Group A and B) each of 30 patients. Group A will be subdivided into 2 groups (1 and 2). All LSC lesions will be treated in any patient having multiple lesions.

* Group 1 - A: Patients will receive 3 monthly laser sessions, in addition to the use of topical emollients only once daily in between the sessions.
* Group 2 - A: Patients will receive 3 monthly laser sessions, in addition to topical steroids twice daily and topical emollient once daily in between the sessions.
* Group B: Patients will be prescribed topical steroids twice daily and topical emollient once daily for 3 months.

to see if:

1. Pruritus severity scale.
2. Scaling, erythema, lichenification excoriation scores
3. Visual analogue scale.
4. Investigator's Global Assessment.
5. Itching mediators (Interleukin-31, Nerve Growth Factor and Substance P assays (itching mediators)
6. Depression

improve more in which group of patients after treatment.

DETAILED DESCRIPTION:
All the patients were subjected to the following:

I. Before treatment:

A. Consent: An informed written consent will be signed by each patient before enrolment in the study.

B. Detailed history taking :

• Personal history: name, age, sex, skin type, occupation, residence, marital status, and smoking.

* History of present illness: onset, course, duration of disease, precipitating factors and any medications.
* Past history of any associated systemic or dermatological diseases.
* Family history of any dermatological disease e.g. psoriasis, atopic dermatitis,….etc.
* Drug history.

C. Skin biopsy: Two 3 mm punch biopsies will be taken from the lesion from each patient under local anesthesia using (Lidocaine®). One for histopathology to confirm diagnosis of LSC and the other for measuring itching mediators in the lesion before treatment by enzyme-linked immunosorbent assay (ELISA)). Another biopsy will be taken from a non lesional skin from same patient for measuring itching mediators by ELISA. Biopsies for ELISA will be stored at -20 degree celsius in eppendorfs with 3 ml phosphate buffer saline (PBS) added to each eppendorf. Tissue samples with PBS will be homogenized by a grinder, then centrifuged for 20 minutes at 3000 revolutions per minute (rpm) speed, the supernatant will be removed to be added to the ELISA kit wells for Human Interleukin-31, Nerve Growth Factor and Substance P assays (itching mediators)

D. Clinical assessment:

1. Pruritus severity scale.
2. Scaling, erythema, lichenification excoriation scores
3. Visual analogue scale.
4. Investigator's Global Assessment.

   E. Depression assessment: Beck Depression Inventory questionnaire will be used to assess the depression in each patient .

   F. Therapeutic Intervention: Patients will be divided as discussed before. - Topical steroids used will be a moderate potency topical steroid.
   * Fractional carbon dioxide laser sessions for groups A (1 and 2) by laser machine.
   * Parameters of laser session: (Parameters will be adjusted according to skin type, lesion thickness and condition) Power 15 to 20 watt according to skin color. Dwell time 800 to1000 milliseconds. Spacing 600 micrometers. Stack 2

   II. After treatment:

   A. Assessment of biochemical efficacy (measuring itching mediators after treatment): After one month from the last session for group A and after one month from stoppage of steroids for group B, a skin biopsy from the plaque (from a nearby site to the former one) will be taken as discussed before for ELISA.

   B. Assessment of clinical efficacy by scores as discussed before.

   C. Depression assessment: Beck Depression Inventory questionnaire will be repeated.

   D. Assessment of safety:
   * Assessment of side effects of laser and their treatment:

   Erythema, burning sensation, PIH, pruritus and/or pixilation. • Assessment of side effects of topical corticosteroids and their treatment: Atrophy, telangiectasia, hypopigmentation, hypertrichosis, purpura, ulceration, irritation, secondary infection.

   • Assessment of side effects of skin biopsy and their treatment: Bleeding, secondary infection and/or Scarring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LSC with no underlying dermatological disease, not on topical or systemic treatment for at least 4 weeks prior to study.

Exclusion Criteria:

* Pregnant and lactating females.
* Patients who are diagnosed with any systemic disease that can result in generalized pruritus (e.g. hepatic, renal, uncontrolled diabetes mellitus, thyroid,….etc ) from history.
* Patients with contraindications to laser e.g., keloidal tendency, post inflammatory hyperpigmentation (PIH).
* Patients with dermatological disease (e.g. psoriasis, atopic dermatitis, ….etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between 2 groups regarding change in Pruritus severity scale | through study completion, an average of 5months
  Minimum value: 3 , Maximum value: 22 , higher scores mean a worse outcome.
Comparison between 2 groups regarding change in Visual analogue scale | through study completion, an average of 5months
  Minimum value:0 , Maximum value: 10, higher scores mean a worse outcome.
Comparison between 2 groups regarding change in Investigator's Global Assessment. | through study completion, an average of 5months
  Minimum value: 0, Maximum value: 3, higher scores mean a worse outcome.
Comparison between 2 groups regarding change in Scaling score | through study completion, an average of 5months
  Minimum value: 0, Maximum value: 3, higher scores mean a worse outcome.
Comparison between 2 groups regarding change in Erythema score | through study completion, an average of 5months
  Minimum value: 0, Maximum value: 3, higher scores mean a worse outcome.
Comparison between 2 groups regarding change in Lichenification score | through study completion, an average of 5months
  Minimum value: 0, Maximum value: 3, higher scores mean a worse outcome.
Comparison between 2 groups regarding change in Excoriation score | through study completion, an average of 5months
  Minimum value: 0, Maximum value: 3, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
change of depression score in both groups. | through study completion, an average of 5months
  Minimum value: 0, Maximum value: 63, higher scores mean a worse outcome.
change of itching mediators' levels (IL-31, Nerve Growth Factor and substance) between 2 groups | through study completion, an average of 5months
  all will be measured by pg/ml
Comparison of itching mediator's levels in lesional, non-lesional skin and healthy controls | through study completion, an average of 5months
  all will be measured by pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Lobna Alieldin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participants' data that underlie reported results will be shared upon request, after deidentification, for researches who provide a methodologically sound proposal to access data to achieve aims in the approved proposal. This is beginning 3 months up to 12 months after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months up to 12 months after publication.
Access Criteria: Researches who provide a methodologically sound proposal to access data to achieve aims in the approved proposal.

REFERENCES:
- [Derived] Esmat S, Sany I, Alieldin L, Nour Z, Azzazi Y. Fractional Carbon Dioxide Laser for Lichen Simplex Chronicus: A Randomized Controlled Trial. Dermatol Surg. 2025 Aug 6. doi: 10.1097/DSS.0000000000004809. Online ahead of print. PMID 40767880